CLINICAL TRIAL: NCT06080490
Title: Factors Affecting the Tacrolimus Blood Concentration and Its Impact on Transplant-related Outcomes in Pediatric HSCT Recipients: a Single-center Retrospective Study
Brief Title: Tacrolimus Blood Concentration and Transplant-related Outcomes in Pediatric HSCT Recipients
Status: Completed | Type: Observational
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Antonello Di Paolo, M.D., Ph.D., Professor of Pharmacology, University of Pisa
Other Study IDs: GEN/INT 0001973
Record Dates: First submitted 2023-10-06; First posted 2023-10-12 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Graft Vs Host Disease; Transplant Failure; Stem Cell Transplant Complications
Keywords: HSCT; Tacrolimus; GVHD; Pediatric patients
MeSH Terms: conditions — Graft vs Host Disease | interventions — Tacrolimus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: TAC C/D ratio — Pharmacokinetics of TAC according to possible influencing factors
  Other Names: Tacrolimus

SUMMARY:
The goal of this retrospective observational study is to investigate any possible association among tacrolimus (TAC) blood concentrations, clinical efficacy and tolerability.

Therefore, the main questions it aims to answer are:

1. to clarify which variables, how and to what extent influence daily TAC blood concentrations in pediatric allo-hematopoietic stem cell transplantation (HSCT) recipients;
2. to investigate the incidence of graft-versus-host disease (GVHD) and graft failure according to TAC exposure.

Pediatric patients administered TAC to prevent GVHD after an allogeneic bone marrow transplantation.

DETAILED DESCRIPTION:
Patients undergoing allo-HSCT will be recruited at IRCC Burlo Garofolo, collecting demographic and clinical characteristics from electronic medical records in a retrospective manner: age, sex, primary disease, donor type and stem cell source, body weight (BW), white blood cell (WBC) count, platelet count, red blood cell (RBC) counts, hemoglobin (HGB) and hematocrit (HCT) levels, red cell concentrate (RCC) transfusions. Other clinical laboratory data (i.e., liver and kidney function) will be included, as well as concomitant drugs administered to patients after allo-HSCT (i.e, mycophenolate mofetil, steroids, pantoprazole, voriconazole, methotrexate). Data will be collected, validated, and presented according to Good Clinical Practice (GCP) principles to support the statistical analyses and subsequent reporting. Once selected according to predefined inclusion requirements, data will be collected anonymously; an identification code will be assigned to each case. As per GCP, all collected information will be recorded, handled, and stored in a way that allows its accurate reporting, interpretation, and verification with user access restriction, and data will be retrievable by designated personnel only.

Because of the retrospective nature of the present research protocol, all eligible patients will be included in the study population only if their medical and laboratory records will be complete.

Statistical analyses (for descriptive and comparative aims) will be performed stratifying patients by body weight, age, gender, and source of stem cells. Univariate and multivariate tests will be used, together with Kaplan-Meyer tes, Cox proportional hazard model and ROC curve analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age of the patients between 0 and 18 years (pediatric)
* Patients undergoing allogeneic bone marrow transplantation
* Patients' GVHD prophylaxis with tacrolimus
* Signed informed consent

Exclusion Criteria:

* Patients undergoing autologous bone marrow transplantation
* Patients not undergoing GVHD prophylaxis
* Patients undergoing cyclosporin prophylaxis
* Incomplete pharmacokinetic/pharmacodynamic data
* Lack of any informed consent

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients who underwent allo-HSCT procedure between January 2011and December 2022 at IRCC Burlo Garofolo
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2023-09-29 (Actual); Primary Completion 2024-09-29 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
TAC pharmacokinetics | 0-30 days
  Evaluation of factors affecting TAC blood concentration/dose (C/D) ratio

SECONDARY OUTCOMES:
GVHD | 0-180 days
  Evaluation of GVHD in patients according to TAC C/D
Graft failure | 0-180 days
  Evaluation of graft failure in patients according to TAC C/D

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Maximova, MD, Principal Investigator — IRCCS Burlo Garofolo - Trieste - ITALY
Locations (1):
- IRCCS Burlo Garofolo, Trieste, Italy

IPD SHARING:
Plan to Share IPD: Undecided
IPD sharing plan is under evaluation by local IRB

REFERENCES:
- [Result] Braidotti S, Curci D, Maestro A, Zanon D, Maximova N, Di Paolo A. Effect of early post-hematopoietic stem cell transplant tacrolimus concentration on transplant outcomes in pediatric recipients: One facility's ten-year experience of immunosuppression with tacrolimus. Int Immunopharmacol. 2024 Sep 10;138:112636. doi: 10.1016/j.intimp.2024.112636. Epub 2024 Jul 10. PMID 38991629